CLINICAL TRIAL: NCT03519074
Title: Phase II Trial of Cisplatin Combined with Oral TS-1 in Patients with Advanced Solid Tumors with Different Degrees of Liver Dysfunction
Brief Title: Cisplatin Combined with Oral TS-1 in Patients with Advanced Solid Tumors with Different Degrees of Liver Dysfunction
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016/00691
Record Dates: First submitted 2018-04-02; First posted 2018-05-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cancer; Liver Dysfunction
MeSH Terms: conditions — Neoplasms; Liver Diseases | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TS-1 combined with cisplatin (Experimental): Eligible patients will be stratified by degree of liver dysfunction into 4 cohorts, in accordance to the National Cancer Institute Organ Dysfunction Working Group (NCI-ODWG) criteria
  Interventions: Drug: TS-1 combined with cisplatin

INTERVENTIONS:
Drug: TS-1 combined with cisplatin — Cisplatin 60mg/m2, day 1, every 21 days Oral TS-1 30mg/m2 bd, days 1-14, every 21 days (absolute dose of oral TS-1 will be 40-60mg bd days 1-14, every 21 days, depending on body surface area)

SUMMARY:
The purpose of this study is to formally characterize the pharmacokinetics (PK), safety, and tolerability of TS-1 in combination with cisplatin in adult patients with advanced solid tumors who have mild, moderate or severe hepatic impairment relative to patients with normal hepatic function, as categorized by the United States National Cancer Institute organ dysfunction working group [NCI-ODWG] criteria for hepatic dysfunction.

DETAILED DESCRIPTION:
Hepatic impairment is a common co-morbidity in cancer patients, particularly in those with extensive liver metastases. Decreased drug clearance as a result of impaired liver function may lead to increased systemic exposure and possibly greater toxicity. As many chemotherapeutic agents are metabolized by the liver, treatment options tend to be limited in patients with severe hepatic impairment, even in the presence of good performance status and adequate other organ function. Cisplatin is an active chemotherapeutic agent with broad spectrum activity that can safely be administered in severe hepatic impairment. Cisplatin has been combined safely with full dose oral TS-1 with good efficacy in a spectrum of solid tumors in patients with adequate renal and hepatic function.

The purpose of this study is to formally characterize the pharmacokinetics (PK), safety, and tolerability of TS-1 in combination with cisplatin in adult patients with advanced solid tumors who have mild, moderate or severe hepatic impairment relative to patients with normal hepatic function, as categorized by the United States National Cancer Institute organ dysfunction working group [NCI-ODWG] criteria for hepatic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

Patients must fulfill ALL the following inclusion criteria

* Age 18 years.
* Histologic or cytologic diagnosis of carcinoma, that is either refractory to standard therapy or has no available therapies.
* Measurable disease using the RECIST v1.1 criteria
* ECOG performance 0 or 1.
* Estimated life expectancy of at least 12 weeks.
* Adequate bone marrow and renal function as follows:

Bone marrow: Absolute neutrophil count (ANC) 1.5 x 109/L Platelets 100 x 109/L Renal: calculated creatinine clearance >60ml/minute Total bilirubin and AST/ALT as described in Table 1

* Able to swallow pills
* Signed informed consent from patient or legal representative
* Patients with reproductive potential must use an approved contraceptive method if appropriate (e.g., intrauterine device, birth control pills, or barrier device) during and for three months after the study.
* Females with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.

Exclusion Criteria:

Patients will be excluded from the study for any of the following reasons:

* Concurrent administration of any other tumor therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Treatment of a small molecule targeted agents ≤ 2 weeks prior to starting study treatment
* Treatment within the last 30 days with any investigational drug.
* Radiotherapy ≤4 weeks prior to starting study treatment or who have not recovered from radiotherapy-related toxicities. Limited field palliative radiotherapy ≤ 2 weeks prior to starting study treatment is allowed
* Major surgery within 28 days of study drug administration.
* History or presence of serious uncontrolled ventricular arrhythmias
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of TS-1 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Known history of human immunodeficiency virus (HIV) seropositivity (HIV testing is not mandatory)
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Pregnancy.
* Breast feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Poorly controlled diabetes mellitus.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment
* Symptomatic brain metastasis.
* History of significant neurological or mental disorder, including seizures or dementia.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-07-22 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Efficacy evaluations: Disease status | Radiological evaluation of tumor status every 2 cycles of cisplatin and oral TS-1 from baseline until documented disease progression; assessed up to 12 months
  Efficacy evaluations will be performed using the RECIST v1.1 criteria
  Measurable disease:
  Tumor lesions: Must be accurately measured in at least one dimension (longest diameter in the plane of measurement is to be recorded) with a minimum size of 10mm on CT scan Malignant lymph node: ≥15mm in short axis on CT scan
  Non-measurable disease: All other lesions, including small lesions (longest diameter <10mm or pathological lymph nodes with >10 to <15mm short axis) as well as truly non-measurable lesions
Efficacy Evaluation: Timing | 5 years
  The duration of tumor response is measured from the date of enrollment until the first date of documented disease progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore, Singapore
  - Ng Teng Fong General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schoffski P. The modulated oral fluoropyrimidine prodrug S-1, and its use in gastrointestinal cancer and other solid tumors. Anticancer Drugs. 2004 Feb;15(2):85-106. doi: 10.1097/00001813-200402000-00001. PMID 15075664
- [Background] Yamamoto D, Iwase S, Tsubota Y, Ariyoshi K, Kawaguchi T, Miyaji T, Sueoka N, Yamamoto C, Teramoto S, Odagiri H, Kitamura K, Nagumo Y, Yamaguchi T. Randomized study of orally administered fluorinated pyrimidines (capecitabine versus S-1) in women with metastatic or recurrent breast cancer: Japan Breast Cancer Research Network 05 Trial. Cancer Chemother Pharmacol. 2015 Jun;75(6):1183-9. doi: 10.1007/s00280-015-2738-3. Epub 2015 Apr 11. PMID 25862350
- [Background] Takashima T, Mukai H, Hara F, Matsubara N, Saito T, Takano T, Park Y, Toyama T, Hozumi Y, Tsurutani J, Imoto S, Watanabe T, Sagara Y, Nishimura R, Shimozuma K, Ohashi Y; SELECT BC Study Group. Taxanes versus S-1 as the first-line chemotherapy for metastatic breast cancer (SELECT BC): an open-label, non-inferiority, randomised phase 3 trial. Lancet Oncol. 2016 Jan;17(1):90-8. doi: 10.1016/S1470-2045(15)00411-8. Epub 2015 Nov 27. PMID 26617202